CLINICAL TRIAL: NCT05738759
Title: Comparative Outcomes of Intraoperative Epidural Application of Anesthetic Cocktail Following Endoscopic Lumbar Discectomy: A Randomized Controlled Trial
Brief Title: RCT - Epidural Anesthetic Cocktail Following Endoscopic Lumbar Discectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 013/2565
Record Dates: First submitted 2022-08-21; First posted 2023-02-22 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Patients were divided into two groups using computer-generated block-of-four randomization. The experimental group received epidural anesthetic cocktail following endoscopic discectomy, while the control group received placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural Anesthetic Cocktail (Experimental): Patients which received epidural anesthetic cocktail following endoscopic discectomy
  Interventions: Drug: Epidural Anesthetic Cocktail
- Placebo (Placebo Comparator): Patients which received placebo following endoscopic discectomy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epidural Anesthetic Cocktail — The anesthetic cocktail, consists of triamcinolone 40 mg, marcaine 5 mg, and morphine 3 mg, is soaked in the gelfoam size 1x2 cm and applied on the epidura before removal of the endoscope.
  Other Names: Cocktail
  Arms: Epidural Anesthetic Cocktail
Drug: Placebo — The placebo is soaked with NSS in the gelfoam size 1x2 cm as well and applied on the epidura before removal of the endoscope.
  Arms: Placebo

SUMMARY:
The study aims to study the effect of intraoperative epidural application of anesthetic cocktail following endoscopic lumbar discectomy in improving postoperative pain, length of hospital stay, time at first dose analgesia, post-operative opioid consumption, functional outcomes, time return to work, and postoperative complications

DETAILED DESCRIPTION:
This is a randomized controlled trial study the effects of epidural anesthetic cocktail. The cocktail, consists of triamcinolone 40 mg, marcaine 5 mg, and morphine 3 mg, is soaked in the gelfoam size 1x2 cm and applied on the epidura before removal of the endoscope. 54 participants are deivided into two arms, experimental and placebo group, and randomized into the trial. Primary objective is the ODI score from patient-reported function outcome at 3 months with secondary objective as mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Lumbar radiculopathy
* No prior spinal surgery or recurrent lumbar disc herniation
* Plan for endoscopic discectomy after failed conservative for at least 6 weeks
* Single-level herniation confirmed by MRI which correlated with symptoms

Exclusion Criteria:

* Allergic or contraindicated to amide-type anesthesia, opioid, NSAIDs, or steroids
* Cauda equina syndrome
* Concomitant with other abnormalities
* Unable to answer questionnaires
* Cannot tolerate surgery due to medical comorbidities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 3rd month
  To compare efficacy of patient-reported functional outcomes achieved with epidural cocktail, measured as Oswestry Disability Index (ODI) at 3 months

SECONDARY OUTCOMES:
Functional Outcomes | POD 1st day, 1st wk, 6th wk, 3th mo, 6th mo, 1st yr
  ODI, VAS of leg pain, VAS of back pain, Modified Macnab score
Postoperative outcomes | POD 1st day, 1st wk, 6th wk, 3th mo, 6th mo, 1st yr
  Time at first dose analgesia, Post-op opioid consumption, complication, time return to work

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Savang Vadhana Memorial Hospital, Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data was save in form of microsoft excel spreadsheet and SPSS file

REFERENCES:
- [Background] Jordan J, Konstantinou K, O'Dowd J. Herniated lumbar disc. BMJ Clin Evid. 2009 Mar 26;2009:1118. PMID 19445754
- [Background] Wilder DG, Pope MH, Frymoyer JW. The biomechanics of lumbar disc herniation and the effect of overload and instability. J Spinal Disord. 1988;1(1):16-32. PMID 2980059
- [Background] Bajwa SJ, Haldar R. Pain management following spinal surgeries: An appraisal of the available options. J Craniovertebr Junction Spine. 2015 Jul-Sep;6(3):105-10. doi: 10.4103/0974-8237.161589. PMID 26288544
- [Background] Sinatra RS, Torres J, Bustos AM. Pain management after major orthopaedic surgery: current strategies and new concepts. J Am Acad Orthop Surg. 2002 Mar-Apr;10(2):117-29. doi: 10.5435/00124635-200203000-00007. PMID 11929206
- [Background] Elder JB, Hoh DJ, Wang MY. Postoperative continuous paravertebral anesthetic infusion for pain control in lumbar spinal fusion surgery. Spine (Phila Pa 1976). 2008 Jan 15;33(2):210-8. doi: 10.1097/BRS.0b013e318160447a. PMID 18197109
- [Background] Jirarattanaphochai K, Jung S, Thienthong S, Krisanaprakornkit W, Sumananont C. Peridural methylprednisolone and wound infiltration with bupivacaine for postoperative pain control after posterior lumbar spine surgery: a randomized double-blinded placebo-controlled trial. Spine (Phila Pa 1976). 2007 Mar 15;32(6):609-16; discussion 617. doi: 10.1097/01.brs.0000257541.91728.a1. PMID 17413463
- [Background] Mirzai H, Tekin I, Alincak H. Perioperative use of corticosteroid and bupivacaine combination in lumbar disc surgery: a randomized controlled trial. Spine (Phila Pa 1976). 2002 Feb 15;27(4):343-6. doi: 10.1097/00007632-200202150-00003. PMID 11840097
- [Background] Du JP, Fan Y, Hao DJ, Huang YF, Zhang JN, Yuan LH. Application of Gelatin Sponge Impregnated with a Mixture of 3 Drugs to Intraoperative Nerve Root Block to Promote Early Postoperative Recovery of Lumbar Disc Herniation. World Neurosurg. 2018 Jun;114:e1168-e1173. doi: 10.1016/j.wneu.2018.03.170. Epub 2018 Mar 31. PMID 29614356
- [Background] Keorochana G, Pairuchvej S, Setrkraising K, Arirachakaran A, Kongtharvonskul J. Comparative Outcomes of Perioperative Epidural Steroids After Percutaneous Endoscopic Lumbar Discectomy for Lumbar Disc Herniation: A Randomized Placebo-Controlled Trial. World Neurosurg. 2018 Nov;119:e244-e249. doi: 10.1016/j.wneu.2018.07.122. Epub 2018 Jul 27. PMID 30059778
- [Background] Kjaergaard M, Moiniche S, Olsen KS. Wound infiltration with local anesthetics for post-operative pain relief in lumbar spine surgery: a systematic review. Acta Anaesthesiol Scand. 2012 Mar;56(3):282-90. doi: 10.1111/j.1399-6576.2011.02629.x. Epub 2012 Jan 19. PMID 22260370
- [Background] Li K, Ji C, Luo D, Feng H, Yang K, Xu H. Wound infiltration with ropivacaine as an adjuvant to patient controlled analgesia for transforaminal lumbar interbody fusion: a retrospective study. BMC Anesthesiol. 2020 Nov 18;20(1):288. doi: 10.1186/s12871-020-01205-5. PMID 33208089
- [Background] Steel T, Jones R, Crossman J, Sheehy J, Bentivoglio P, Pell M. Intraoperative wound infiltration with bupivacaine in patients undergoing lumbar spine surgery. J Clin Neurosci. 1998 Jul;5(3):298-303. doi: 10.1016/s0967-5868(98)90065-0. PMID 18639036
- [Background] Ersayli DT, Gurbet A, Bekar A, Uckunkaya N, Bilgin H. Effects of perioperatively administered bupivacaine and bupivacaine-methylprednisolone on pain after lumbar discectomy. Spine (Phila Pa 1976). 2006 Sep 1;31(19):2221-6. doi: 10.1097/01.brs.0000232801.19965.a0. PMID 16946657
- [Background] Arirachakaran A, Siripaiboonkij M, Pairuchvej S, Setrkraising K, Pruttikul P, Piyasakulkaew C, Kongtharvonskul J. Comparative outcomes of epidural steroids versus placebo after lumbar discectomy in lumbar disc herniation: a systematic review and meta-analysis of randomized controlled trials. Eur J Orthop Surg Traumatol. 2018 Dec;28(8):1589-1599. doi: 10.1007/s00590-018-2229-4. Epub 2018 May 29. PMID 29845327
- [Background] Jamjoom BA, Jamjoom AB. Efficacy of intraoperative epidural steroids in lumbar discectomy: a systematic review. BMC Musculoskelet Disord. 2014 May 5;15:146. doi: 10.1186/1471-2474-15-146. PMID 24885519
- [Background] Wilson-Smith A, Chang N, Lu VM, Mobbs RJ, Fadhil M, Lloyd D, Kim S, Phan K. Epidural Steroids at Closure After Microdiscectomy/Laminectomy for Reduction of Postoperative Analgesia: Systematic Review and Meta-Analysis. World Neurosurg. 2018 Feb;110:e212-e221. doi: 10.1016/j.wneu.2017.10.133. Epub 2017 Nov 1. PMID 29102751
- [Background] Akinduro OO, Miller BA, Haussen DC, Pradilla G, Ahmad FU. Complications of intraoperative epidural steroid use in lumbar discectomy: a systematic review and meta-analysis. Neurosurg Focus. 2015 Oct;39(4):E12. doi: 10.3171/2015.7.FOCUS15269. PMID 26424336
- [Background] McNeill TW, Andersson GB, Schell B, Sinkora G, Nelson J, Lavender SA. Epidural administration of methylprednisolone and morphine for pain after a spinal operation. A randomized, prospective, comparative study. J Bone Joint Surg Am. 1995 Dec;77(12):1814-8. doi: 10.2106/00004623-199512000-00004. PMID 8550648
- [Background] Bahari S, El-Dahab M, Cleary M, Sparkes J. Efficacy of triamcinolone acetonide and bupivacaine for pain after lumbar discectomy. Eur Spine J. 2010 Jul;19(7):1099-103. doi: 10.1007/s00586-010-1360-7. Epub 2010 Mar 12. PMID 20224868
- [Background] Samoladas E, Kapinas A, Papadopoulos DV, Gkiatas I, Papastefanou S, Gelalis ID. Intraoperative epidural application of steroid and local anaesthetic agent following lumbar discectomy: A prospective double blinded randomized controlled trial. J Clin Orthop Trauma. 2019 Oct;10(Suppl 1):S143-S146. doi: 10.1016/j.jcot.2019.03.005. Epub 2019 Mar 12. PMID 31695273
- [Background] Copay AG, Glassman SD, Subach BR, Berven S, Schuler TC, Carreon LY. Minimum clinically important difference in lumbar spine surgery patients: a choice of methods using the Oswestry Disability Index, Medical Outcomes Study questionnaire Short Form 36, and pain scales. Spine J. 2008 Nov-Dec;8(6):968-74. doi: 10.1016/j.spinee.2007.11.006. Epub 2008 Jan 16. PMID 18201937